CLINICAL TRIAL: NCT06424457
Title: Video Assisted Thoracoscopic Surgery (VATS) Versus Thoracotomy in Management of Empyema in Pediatric Patients
Brief Title: Pediatric Video Assisted Thoracoscopic Surgery (VATS) in Management of Empyema
Acronym: VATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali zein elabdein abd elaleim, Principal investigator, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 04-2024-100227
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Thoracic Empyema
Keywords: pediatric empyema; VATS decortication
MeSH Terms: conditions — Empyema, Pleural | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (VATS) (Experimental): (group A) will receive VATS decortication as their definite management
  Interventions: Procedure: video assisted thoracoscopy (VATS)
- group B (open thoracotomy) (Experimental): (group B) will be assigned to open thoracotomy
  Interventions: Procedure: open thoracotomy

INTERVENTIONS:
Procedure: video assisted thoracoscopy (VATS) — the investigators compare the outcomes of intervention by VATS and doing complete decortication or open surgery thoracotomy
  Arms: group A (VATS)
Procedure: open thoracotomy — the investigators assess the outcomes of intervention by doing complete decortication through open surgery thoracotomy
  Arms: group B (open thoracotomy)

SUMMARY:
Thoracic surgeons have developed a thoracoscopic procedure which is less intrusive method allows complete evacuation and washing of the debris from the pleural cavity. This approach may also have the benefit of less invasive maneuver, a shorter hospital stay and a decreased rate of postoperative complications.

The aim of this study is to evaluate the advantages and disadvantages of the video-assisted thoracoscopic surgery (VATS) approach in comparison with thoracotomy in management of empyema in pediatric patients.

DETAILED DESCRIPTION:
comparison between VATS decortication and open thoracotomy in cases of pediatric empyema

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients 1 yrs. : ≤ 18 yrs.
* Patients with empyema due to pneumonia.
* Patients with empyema had lasted for fewer than 3 weeks.

Exclusion Criteria:

* Patients < 1 yrs. old.
* Patients with whom pleural empyema had lasted for more than 3 weeks.
* Patients with empyema had been caused by trauma.
* Patients whose parents refuse to be included in the study.
* Patients with empyema due to ruptured lung abscess.
* Patients with empyema due to chest wall abscess.
* Patients with empyema due to rib osteomyelitis.
* Patients with bronchopleural fistula.
* Patients with post-surgical empyema.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
wound size | after 1week post operative
  by centimeters
wound infection | during 1week post operative
  which degree of infection or if there is a burst wound
hospital stay | 1week post operative
  by days post operative
air leak duration | during 1week post operative
  by days and takes how many days to stop air leakage
pain score | during 1week post operative.
  through pain score scale 0 No Pain 1-3 Mild Pain (nagging, annoying) 4-6 Moderate Pain 7-10 Severe Pain (disabling)
Early mobilization. | during 1week post operative
  how many days

SECONDARY OUTCOMES:
chronic pain | after 1month post operative
  presented or not
avoidance of scoliosis | after 1month post operative
  which degree
shoulder muscle girdle weakness and deformity. | after 1month post operative
  yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ayyad, prof., Study Director — professor; Mahmoud sallam, MD, Study Director — doctor
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold DT, Hamilton FW, Morris TT, Suri T, Morley A, Frost V, Vipond IB, Medford AR, Payne RA, Muir P, Maskell NA. Epidemiology of pleural empyema in English hospitals and the impact of influenza. Eur Respir J. 2021 Jun 17;57(6):2003546. doi: 10.1183/13993003.03546-2020. Print 2021 Jun. PMID 33334937
- [Background] Krenke K, Urbankowska E, Urbankowski T, Lange J, Kulus M. Clinical characteristics of 323 children with parapneumonic pleural effusion and pleural empyema due to community acquired pneumonia. J Infect Chemother. 2016 May;22(5):292-7. doi: 10.1016/j.jiac.2016.01.016. Epub 2016 Feb 23. PMID 26919911
- [Background] Shojaee S, Lee HJ. Thoracoscopy: medical versus surgical-in the management of pleural diseases. J Thorac Dis. 2015 Dec;7(Suppl 4):S339-51. doi: 10.3978/j.issn.2072-1439.2015.11.66. PMID 26807282
- [Background] Bedawi EO, Hassan M, McCracken D, Rahman NM. Pleural infection: a closer look at the etiopathogenesis, microbiology and role of antibiotics. Expert Rev Respir Med. 2019 Apr;13(4):337-347. doi: 10.1080/17476348.2019.1578212. Epub 2019 Feb 20. PMID 30707629